CLINICAL TRIAL: NCT01573598
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Relapse Prevention Study With Vilazodone in Patients With Major Depressive Disorder
Brief Title: Safety and Efficacy of Vilazodone in Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VLZ-MD-02
Record Dates: First submitted 2012-04-04; First posted 2012-04-09 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Vilazodone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Dose-matched placebo capsules, oral administration
  Interventions: Drug: Placebo
- Vilazodone 20mg (Experimental): Vilazodone tablets, 20 mg per day, oral administration
  Interventions: Drug: Vilazodone
- Vilazodone 40mg (Experimental): Vilazodone tablets, 40 mg per day, oral administration
  Interventions: Drug: Vilazodone

INTERVENTIONS:
Drug: Placebo — Matching placebo given orally, once per day
  Arms: Placebo
Drug: Vilazodone — Vilazodone, 20 mg per day, oral administration
  Other Names: Viibryd
  Arms: Vilazodone 20mg
Drug: Vilazodone — Vilazodone, 40 mg once per day, oral administration
  Other Names: Viibryd
  Arms: Vilazodone 40mg

SUMMARY:
Safety and Efficacy of Vilazodone in Major Depressive Disorder

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-70 years of age
* Currently meet the DSM-IV-TR criteria for Major Depressive Disorder
* The patient's current major depressive episode must be at least 8 weeks and no longer than 18 months in duration

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women of childbearing potential who are not practicing a reliable method of birth control
* Patients with a history of meeting DSM-IV-TR criteria for:

  * any manic, hypomanic or mixed episode, including bipolar disorder and substance-induced manic, hypomanic, or mixed episode;
  * any depressive episode with psychotic or catatonic features;
  * panic disorder with or without agoraphobia;
  * obsessive-compulsive disorder;
  * Schizophrenia, schizoaffective, or other psychotic disorder;
  * bulimia or anorexia nervosa;
  * presence of borderline personality disorder or antisocial personality disorder; h. mental retardation, dementia, amnesia, or other cognitive disorders
* Patients who are considered a suicide risk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1219 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Time to first relapse during the double-blind treatment phase | Number of days from the randomization date to the relapse date, up to 28 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Reichley, Study Director — Forest Research Institute, a subsidiary of Actavis plc.
Locations (75):
- United States (38):
  - Forest Investigative Site 030, Beverly Hills, California
  - Forest Investigative Site 012, Chino, California
  - Forest Investigative Site 022, Costa Mesa, California
  - Forest Investigative Site 017, Los Angeles, California
  - Forest Investigative Site 005, Newport Beach, California
  - Forest Investigative Site 027, Riverside, California
  - Forest Investigative Site 026, San Diego, California
  - Forest Investigative Site 016, Cromwell, Connecticut
  - Forest Investigative Site 029, Hartford, Connecticut
  - Forest Investigative Site 020, Doral, Florida
  - Forest Investigative Site 007, Fort Lauderdale, Florida
  - Forest Investigative Site 006, Fort Myers, Florida
  - Forest Investigative Site 004, Hallandale, Florida
  - Forest Investigative Site 039, Jacksonville, Florida
  - Forest Investigative Site 008, Jacksonville Beach, Florida
  - Forest Investigative Site 015, Leesburg, Florida
  - Forest Investigative Site 035, Orlando, Florida
  - Forest Investigative Site 001, West Palm Beach, Florida
  - Forest Investigative Site 034, Winter Park, Florida
  - Forest Investigative Site 019, Hoffman Estates, Illinois
  - Forest Investigative Site 021, Indianapolis, Indiana
  - Forest Investigative Site 003, Boston, Massachusetts
  - Forest Investigative Site 013, Weymouth, Massachusetts
  - Forest Investigative Site 028, Rochester Hills, Michigan
  - Forest Investigative Site 038, Brooklyn, New York
  - Forest Investigative Site 037, New York, New York
  - Forest Investigative Site 032, New York, New York
  - Forest Investigative Site 009, New York, New York
  - Forest Investigative Site 014, Durham, North Carolina
  - Forest Investigative Site 025, Oklahoma City, Oklahoma
  - Forest Investigative Site 024, Oklahoma City, Oklahoma
  - Forest Investigative Site 036, Memphis, Tennessee
  - Forest Investigative Site 023, Dallas, Texas
  - Forest Investigative Site 011, Houston, Texas
  - Forest Investigative Site 010, Plano, Texas
  - Forest Investigative Site 002, San Antonio, Texas
  - Forest Investigative Site 031, Richmond, Virginia
  - Forest Investigative Site 033, Bellevue, Washington
- Bulgaria (4):
  - Forest Investigative Site 103, Pleven
  - Forest Investigative Site 104, Plovdiv
  - Forest Investigative Site 106, Sofia
  - Forest Investigative Site 102, Sofia
- Finland (7):
  - Forest Investigative Site 304, Helsinki, Etelä-Suomen Lääni
  - Forest Investigative Site 305, Helsinki, Etelä-Suomen Lääni
  - Forest Investigative Site 301, Helsinki, Etelä-Suomen Lääni
  - Forest Investigative Site 303, Rauma, Länsi-Suomen Lääni
  - Forest Investigative Site 302, Kuopio
  - Forest Investigative Site 306, Turku
  - Forest Investigative Site 307, Turku
- Germany (9):
  - Forest Investigative Site 401, Hanover, Lower Saxony
  - Forest Investigative Site 405, Dresden, Saxony
  - Forest Investigative Site 403, Berlin
  - Forest Investigative Site 408, Berlin
  - Forest Investigative Site 407, Chemnitz
  - Forest Investigative Site 402, Hüttenberg
  - Forest Investigative Site 409, Münster
  - Forest Investigative Site 404, Nuremberg
  - Forest Investigative Site 406, Westerstede
- Romania (3):
  - Forest Investigative Site 602, Bucharest, București
  - Forest Investigative Site 601, Arad
  - Forest Investigative Site 603, Iași
- Russia (2):
  - Forest Investigative Site 705, Petrozavodsk, Kareliya, Respublika
  - Forest Investigative Site 701, Moscow
- Serbia (6):
  - Forest Investigative Site 804, Belgrade, Beograd
  - Forest Investigative Site 806, Niš, Nišava
  - Forest Investigative Site 801, Belgrade
  - Forest Investigative Site 802, Belgrade
  - Forest Investigative Site 803, Kragujevac
  - Forest Investigative Site 805, Kragujevac, Šumadija
- Ukraine (6):
  - Forest Investigative Site 903, Kherson, Kherson Oblast
  - Forest Investigative Site 905, Luhansk, Luhansk Oblast
  - Forest Investigative Site 901, Lviv, Lviv Oblast
  - Forest Investigative Site 906, Odesa, Odesa Oblast
  - Forest Investigative Site 902, Dnipropetrovsk
  - Forest Investigative Site 904, Simferopol